CLINICAL TRIAL: NCT00734799
Title: Treating Co-Morbid Sleep Difficulties in Veterans With PTSD: A Pilot Study
Brief Title: Treating Co-Morbid Sleep Difficulties in Veterans With Posttraumatic Stress Disorder (PTSD): A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christi Ulmer, Clinical Research Psychologist, Durham VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMR01252
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Posttraumatic Stress Disorder; Insomnia
Keywords: Posttraumatic Stress Disorder; Insomnia,; Imagery Rehearsal Therapy,; IRT,; Cognitive Behavioral Therapy for Insomnia,; CBTI.
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Usual Care/Wait-List Control
- 1 (Experimental): Sleep Intervention for PTSD (SIP)
  Interventions: Behavioral: Sleep Intervention for PTSD (SIP).

INTERVENTIONS:
Behavioral: Sleep Intervention for PTSD (SIP). — Patients in the SIP condition will receive the same elements as the Usual Care patients. In addition, these patients will receive six, bi-weekly, 1-hour individual sessions with the PI, including 3 sessions of Cognitive-Behavioral Therapy for Insomnia (CBT-I) and 3 sessions of Imagery Rehearsal Therapy (IRT). CBT-I consists of education designed to correct unrealistic sleep expectations, a prescription for an individually-tailored behavioral regimen, standard sleep hygiene recommendations, and the identification and restructuring of dysfunctional beliefs and attitudes regarding sleep. IRT is a brief intervention designed to facilitate the patient's "rescripting" of reoccurring nightmares to decrease their associated affective distress.
  Arms: 1

SUMMARY:
A substantial number of US Veterans are suffering from Posttraumatic Stress Disorder (PTSD) following deployment in recent military conflicts, and sleep disturbance is a primary complaint of Veterans presenting to the VA with PTSD. Veterans with PTSD have more self-reported and physician-rated health problems, and health status is associated with PTSD symptom severity. Most Veterans meeting criteria for PTSD report difficulty initiating or maintaining sleep (70-91%), and increased PTSD severity is associated with increased sleep disturbance. Even after receiving treatment for PTSD, Veterans continue to experience residual insomnia at a rate of about 50%, in spite of having achieved PTSD remission.

There are currently no PTSD-specific sleep interventions available, excepting an intervention that is specific to nightmares. Given the prevalence of sleep disturbance in Veterans with PTSD, the absence of interventions for PTSD-related sleep problems, and the increasing number of post-deployment Veterans with trauma-related sleep difficulties, such interventions are desperately needed. In this study, we will test the effectiveness of a multi-component cognitive-behavioral sleep intervention for PTSD that targets both nightmares and insomnia for improving the overall sleep experience of Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) Veterans with PTSD who are also receiving usual care. The primary objective is to pilot test the intervention for efficacy in reducing sleep disturbance. The secondary objective is to examine the relative impact of the intervention on PTSD symptoms. The project is a prospective, randomized, clinical intervention trial. Participants will be randomly assigned to a multi-component cognitive-behavioral sleep intervention for PTSD + Usual Care, or Usual Care alone. We are hypothesizing that 1) Veterans receiving the sleep intervention plus usual care will produce greater improvements (reduced total wake time, increased sleep efficiency, etc) in subjective sleep measures than will Usual Care alone; 2) Veterans receiving the sleep intervention plus usual care will produce greater improvements in nightmare frequency and severity than will Usual Care alone; and 3) the relationship between PTSD symptoms and treatment group will be significantly related to sleep quality in the period intervening baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria: Participants will be recruited from the population of Operation Iraqi Freedom/Operation Enduring Freedom veterans referred to the Posttraumatic Stress Disorder (PTSD) clinic for evaluation and treatment, and volunteers participating in the Mental Illness Research, Education and Clinical Centers (MIRECC) registry who agreed to be recontacted for future studies. All study participants will have: 1) provided informed consent; 2) utilize Durham VA Medical Center health care services as their primary source of health care; 3) will meet the Diagnostic and Statistical Manual (DSM-IV-R) criteria for a diagnosis of PTSD; 4) will screen positive for an Insomnia Disorder on the Duke Structured Sleep Interview for Sleep Disorders (DSISD); 5) and will score greater than 14 on the Insomnia Severity Index (ISI).

Exclusion Criteria: Patients who screen positive on the DSISD for symptoms of Sleep Apnea, Narcolepsy, Restless Legs Syndrome or Circadian Disorders will be excluded from the study. Participants with active drug or alcohol abuse or dependence will be excluded as well.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christi S Ulmer, PhD, Principal Investigator — Durham VAMC
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Ulmer CS, Edinger JD, Calhoun PS. A multi-component cognitive-behavioral intervention for sleep disturbance in veterans with PTSD: a pilot study. J Clin Sleep Med. 2011 Feb 15;7(1):57-68. PMID 21344046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited between 1/1/2008 and 12/31/2009 using flyers placed throughout the VA hospital and a community Veteran Center, and through letters sent to recently deployed veterans who had enrolled in a VA research registry and who had agreed to be recontacted for participation in VA research.
Pre-assignment Details: Of the 93 self-referred prospective study participants, 22 individuals (15 men and 7 women) met study selection criteria, completed baseline procedures, and were subsequently randomized to treatment conditions.
Groups:
- Wait List: Usual Care/Wait-List Control
- Intervention: Sleep Intervention for PTSD (SIP)
Period: Overall Study
Arm/Group | Wait List | Intervention
Started | 9 | 13
Completed | 9 | 9
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait List | Intervention | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 13 | 21
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.22 (11.62) | 47.00 (9.47) | 48.61 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 22
Insomnia Severity [Mean (Standard Deviation); unit: units on a scale] — The ISI is a 7-item questionnaire that provides a global measure of perceived insomnia severity. Each item is rated on a 5-point Likert scale, and the total score ranges from 0-28. The following guidelines are recommended for interpreting the total score: 0-7 (no clinical insomnia), 8-14 (subthreshold insomnia), 15-21 (insomnia of moderate severity), and 22-28 (severe insomnia). The ISI was used to determine treatment eligibility, to assess treatment outcome, and to determine clinical significance of study findings.
  units on a scale | 22.00 (3.97) | 22.77 (4.57) | 22.46 (4.25)
Sleep Quality [Mean (Standard Deviation); unit: units on a scale] — Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a self-rating scale that yields a quantitative index of general sleep quality/disturbances. The PSQI is composed of 4 open-ended questions and 19 self-rated items (0-3 scale) assessing sleep quality and disturbances over a 1-month interval, and yields aglobal score of sleep quality, ranging from 0 to 21. A PSQI cutoff score of 5 is a sensitive and specific value for predicting both clinical and laboratory assessments of sleep.
  units on a scale | 14.33 (3.35) | 14.17 (3.27) | 14.24 (3.22)
PTSD Symptom Checklist-M [Mean (Standard Deviation); unit: scores on a scale] — The PCL-M is a 17-item self-report measure reflecting the degree to which veterans were bothered by each of 17 DSM-IV symptoms of PTSD in the past month. It is rated on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). The total score can range from 17 to 85, with higher scores reflecting greater PTSD symptomatology. In Vietnam veterans, a PCL-M score ≥ 50 was found to be highly predictive of PTSD diagnosis using the SCID. The PCL-M was used to assess treatment outcome and as an indicator of clinical significance of study findings.
  scores on a scale | 63.44 (11.66) | 63.08 (12.47) | 63.23 (11.86)
Depression [Mean (Standard Deviation); unit: scores on a scale] — Depression was assessed using the PHQ-9. The PHQ-2 is a 2-item depression screening instrument that assesses frequency of depressed mood and anhedonia on a scale of 0 (not at all) to 3 (nearly every day). In a primary care population, the PHQ-2 has a sensitivity of 86% and specificity of 78% for detecting major depression, with a score ≥ 2 correctly categorizing the greatest number of those with major depression.
  scores on a scale | 3.88 (2.08) | 3.77 (1.74) | 3.82 (1.84)
Sleep-Specific PTSD Symptoms [Mean (Standard Deviation); unit: scores on a scale] — The Pittsburgh Sleep Quality Index Addendum for PTSD (PSQIA) was used to assess PTSD-related sleep quality, and has acceptable psychometric properties. A cut-off score of 4 was found to have excellent sensitivity and specificity for discriminating those without PTSD from those with PTSD. Total scores on the PSQIA range from 0 to 21, with higher scores reflecting poorer PTSD-related sleep quality.
  scores on a scale | 10.00 (5.29) | 10.00 (4.10) | 10.00 (4.50)
Nightmare Frequency [Mean (Standard Deviation); unit: Number of nightmares per night] — Nightmare frequency was assessed using an electronic sleep diary. The number and severity of nightmares were obtained using a hand-held computer that was programmed to elicit daily responses from participants and electronically record multiple days of subjective sleep information, in addition to the number and severity of nightmares for the previous night. Nightmare frequency (number of nightmares per night) was one of five variables collected from electronic sleep diaries. The average nightmare frequency per night was calculated over a period of 1 week.
  Number of nightmares per night | 0.59 (0.68) | 0.72 (0.43) | 0.67 (0.53)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity
Description: Insomnia severity was assessed using the Insomnia Severity Index (ISI). The ISI is a 7-item questionnaire that provides a global measure of perceived insomnia severity. Each item is rated on a 5-point Likert scale, and the total score ranges from 0-28. The following guidelines are recommended for interpreting the total score: 0-7 (no clinical insomnia), 8-14 (subthreshold insomnia), 15-21 (insomnia of moderate severity), and 22-28 (severe insomnia). The ISI was used to determine treatment eligibility, to assess treatment outcome, and to determine clinical significance of study findings. Participants were assessed at baseline and following a 12-week intervention period.
Time Frame: 12-weeks after Baseline
Population: Intent to treat and completed were both reported. Data on completers reported here.
Measure: Mean (Standard Error); unit: ISI Score
Arm/Group | Wait List | Intervention
Number analyzed (Participants) | 9 | 9
ISI Score | 21.58 (1.90) | 12.45 (1.90)

2. Secondary Outcome: Nightmare Frequency
Description: Nightmare frequency was assessed using an electronic sleep diary. Diary data was collected for a period of 1 week at both baseline and 12 weeks after baseline. The number and severity of nightmares over a 1-week period were obtained using a hand-held computer (PDA) containing an interactive program that automates the collection of subjective sleep data. The PDA device was programmed to elicit daily responses from participants and electronically record multiple days of subjective sleep information, in addition to the number and severity of nightmares for the previous night. Nightmare frequency (number of nightmares per night) was one of five variables collected from electronic sleep diaries.
Time Frame: 12 weeks after Baseline
Measure: Mean (Standard Error); unit: Nightmare frequency per night
Arm/Group | Wait List | Intervention
Number analyzed (Participants) | 9 | 9
Nightmare frequency per night | 0.83 (0.17) | 0.51 (0.18)

ADVERSE EVENTS:
Arm/Group | Wait List | Intervention
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/9 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No